CLINICAL TRIAL: NCT07298980
Title: Expressive Writing in Breast Cancer - The ExBRAC Trial
Brief Title: ExBRAC- Expressive Writing in Breast Cancer
Acronym: ExBRAC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023-2888
Record Dates: First submitted 2025-09-18; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; quality of life; expressive writing
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Writing (Experimental): Expressive writing for 20 minutes, once a week, for 4 consecutive weeks. The intervention is done in addition to standard care.
  Interventions: Behavioral: Expressive Writing
- Control group (No Intervention): No intervention. Treatment according to standard care.

INTERVENTIONS:
Behavioral: Expressive Writing — Expressive writing means that the patient writes privately about the cancer or other related subject for 20 minutes. This will be repeated once a week for 4 weeks. The writing should be done in a place free from distractions and on the patients' mother tongue. The text will not be collected.
  Arms: Expressive Writing

SUMMARY:
The study is a randomized trial designed to examine whether an "expressive writing" intervention can affect the quality of life in patients recently diagnosed with breast cancer. The method "expressive writing" consists of writing about the breast cancer or other related subjects during 20 minutes, once a week for four consecutive weeks. The impact on quality of life will be assessed by having participants complete questionnaires at three different time points during the study. The questionnaire will be developed using a clinimetric approach, based on semi-structured interviews with breast cancer patients. The themes emerging from these interviews will be used to formulate the questions. Additionally, well-known quality-of-life measurement instruments and registry data with clinically relevant information-such as tumor stage and treatment-will be incorporated.

ELIGIBILITY:
Inclusion Criteria:

* Planned for surgery of breast cancer without neoadjuvant treatment

Exclusion Criteria:

* Not able to understand Swedish
* Previous breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | At the 12 months follow-up
  According to EQ-5D-5L VAS. The scale ranges from 0-100 where 0 is "worst possible health" and 100 is "best possible health".

CONTACTS AND LOCATIONS:
Overall Officials: Linnea Huss, M.D., Ph.D., Principal Investigator — Lund University
Locations (1):
- Department of Surgery, Hospital of Helsingborg, Helsingborg, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The ExBRAC Pilot Study — https://clinicaltrials.gov/study/NCT06230068?term=exbrac&rank=1